CLINICAL TRIAL: NCT04704791
Title: Surgical PA-LAA Shunting for Management of Systemic Embolization in Patients With Atrial Fibrillation: a Feasibility Study
Brief Title: Surgical PA-LAA Shunting: a Feasibility Study
Acronym: PA-LAA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to enroll
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Benjamin Hibbert, MD, MD PhD FRCPC Interventional Cardiologist, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20200646-01H
Record Dates: First submitted 2020-11-02; First posted 2021-01-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: LAA Thrombus Prevention
Keywords: shunting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedure arm (Experimental): At the time of surgery a covered stent will be inserted through the atriotomy into the left pulmonary artery and balloon dilated to stabilize the device. The target shunt diameter will be 3.5-4 mm to minimize LAA stasis.
  Interventions: Procedure: PA-LAA shunt

INTERVENTIONS:
Procedure: PA-LAA shunt — At the time of surgery a covered stent will be inserted through the atriotomy into the left pulmonary artery and balloon dilated to stabilize the device. The target shunt diameter will be 3.5-4 mm to minimize LAA stasis.

SUMMARY:
Atrial fibrillation is common and increases the risk of stroke. Traditionally patients are treated with blood thinning medications or at the time of surgery the part of the heart where blood clots form is cut out. Surgically cutting out the left atrial appendage can be difficult and complications can occur. An alternative strategy is to create a tunnel to increase blood flow and wash out the part of the heart where clots form.

This strategy has not been previously studied. The purpose of this study is to determine if creating a tunnel to increase blood flow is feasible and safe.

DETAILED DESCRIPTION:
The goal is to understand the potential avenues to increase Left Atrial Appendage (LAA) flow in patients with Atrial Fibrillation (AF) to minimize systemic embolization risk. Flow modeling demonstrates that the anatomy of the LAA results in decreased velocities in the LAA apex. Introduction of a 3-4mm shunt in the apex can result in increased velocity, less stasis and a lower propensity for thrombus formation. Small (<8mm) inter-chamber shunts can exist in humans with no long term hemodynamic consequences in otherwise structurally normal hearts - making a strategy of pulmonary artery (PA) to LAA shunt an attractive potential therapy given anatomic proximity and gradient differential between the cardiac chambers.

This will be a 5 patient first-in-human feasibility study. The population will include patients undergoing CABG or other cardiovascular surgery with AF and a CHADS2 score >1 in whom the treating team deems traditional therapy with anticoagulants is prohibitive or ineffective (dialysis or EGFR preoperatively <15, previous bleeding with non-reversible pathology, clinically deemed contraindicated to oral anticoagulant). The intervention will be PA-LAA shunt creation at the time of surgery. As this is a single arm study there will be no comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years undergoing CV surgery
* History of AF with a CHADS2 score >1
* Relative contraindication to OAC as determined by the heart team

  1. Dialysis or preoperative eGFR of <15
  2. Bleeding on DOAC/Coumadin with non-reversible pathology
  3. Other medical condition that makes the patient ineligible for OAC
* Anatomic proximity of LAA and PA on preoperative CT scan suitable for shunt creation

Exclusion Criteria:

* LVEF <40%
* History of VTE - either DVT or PE
* Resting baseline preoperative O2 sats <98%
* Inability of the patient to provide written informed consent
* Greater than moderate valvular heart disease which is not to be addressed during surgical intervention
* Documented mPA to PCWP <5mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Composite of device safety and performance | 3 months
  At three months feasibility will be met if there is no:
  1. Device related complications
     1. Bleeding attributable to device implantation
     2. Reintervention (surgical or percutaneous) on the shunt
     3. Resting systemic saturations <92%
     4. Documented Qp:Qs <0.8
  2. Device related performance a. Shunt patency at 3 months as assessed by TEE

SECONDARY OUTCOMES:
Device related performance - maintaining patency | 1 year
  Shunt patency as assessed by TEE
Systemic embolization | 1 year
  Systemic embolization - includes stroke, TIA, MI or peripheral embolization attributable to either LAA thrombus or paradoxical embolization as clinically diagnosed by treating physician
Systemic saturations | 1 year
  Resting saturations <92% - threshold
Need for intervention to close the shunt | 1 year
  Need for intervention to close the shunt either surgically or percutaneously to

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hibbert, MD PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No